CLINICAL TRIAL: NCT06033664
Title: Grocery Prescription Program for Medicaid Adults With Hypertension or Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alison Gustafson (Other)
Collaborators: Instacart Health (Unknown); Kentucky Association of Health Plans (Unknown)
Responsible Party: Sponsor-Investigator, Alison Gustafson, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 88696
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
Keywords: Food Insecurity; Food as Medicine; Medicaid Adults
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Food; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Grocery Prescription Program (Experimental): Participants will receive the Fresh Funds through Instacart
  Interventions: Behavioral: Fresh Funds

INTERVENTIONS:
Behavioral: Fresh Funds — Participants will enroll in Instacart Fresh Funds program. Once enrolled participants will select foods that are eligible in the Fresh Funds to be delivered to their home each week for 12 weeks.
  Other Names: Grocery Prescription Program; Food As Medicine

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a grocery prescription program in adults diagnosed with either Type 2 Diabetes Mellitus or Hypertension. Participants will enroll in Instacart Fresh Funds program. Once enrolled each week participants will select foods that are eligible in the Fresh Funds Program to be delivered to their home for 12 weeks. Participants will also participate in a survey at the beginning of the study and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes Mellitus, hemoglobin A1c = 7.0% and = 12.0% in last 12 months, or diagnosis of hypertension
* Experiencing food insecurity as indicated by 2-item Hunger Vital Sign
* English speaking
* No plans to move from the area for at least 1 year
* Willing and able to accept text messages
* Free living to the extent that participant has control over dietary intake
* Willing and able to provide written informed consent and participate in all study activities.

Exclusion Criteria:

* Participant in diabetes, nutrition, or weight research intervention in last 12 months
* Another member of the household is already enrolled in this study
* Considering bariatric surgery in the next year or prior bariatric surgery
* Lack of safe, stable residence and ability to store meals

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with a percentage change in Hemoglobin A1C (HbgA1C) | baseline and post intervention, approximately 12 weeks
  HbgA1C will be obtained baseline and post intervention by the healthcare provider from the medical chart.

SECONDARY OUTCOMES:
Change in blood pressure | baseline and post intervention, approximately 12 weeks
  Both systolic and diastolic blood pressure will be obtained baseline and post intervention by the healthcare provider from the medical chart.
Change in food insecurity | baseline and post intervention, approximately 12 weeks
  The USDA 6 item food insecurity screener will be used. The scale ranges from 0 to 6 with a higher score indicating greater food insecurity.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Gustafson, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- [Derived] Mayfield C, Lauckner C, Bush J, Cosson E, Batey L, Gustafson A. Development of a statewide network hub for screening, referral, and enrollment into food as medicine programs across Kentucky. Front Public Health. 2025 Jan 7;12:1502858. doi: 10.3389/fpubh.2024.1502858. eCollection 2024. PMID 39845669